CLINICAL TRIAL: NCT07178340
Title: Prospective, Single-arm, Single-center Phase II Clinical Study of Perioperative Therapy for Locally Advanced HER2-negative Hepatoid Adenocarcinoma of Stomach
Brief Title: Perioperative Therapy for HER2-negative Hepatoid Adenocarcinoma of Stomach
Acronym: HASCHANGE02
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LGH2025138
Record Dates: First submitted 2025-09-10; First posted 2025-09-17 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Hepatoid Adenocarcinoma of Stomach
Keywords: HER2; SOX; PD-1 inhibitor; perioperative treatment
MeSH Terms: interventions — Albumin-Bound Paclitaxel; Oxaliplatin; Tegafur; gimeracil; sintilimab

STUDY DESIGN:
Intervention Model Description: perioperative treatment with albumin-bound paclitaxel, oxaliplatin, tegafur,gimeracil and oteracil porassium capsules and sintilimab
Masking Description: Masking Description
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Perioperative treatment for hepatoid adenocarcinoma of stomach (Experimental)
  Interventions: Drug: Perioperative treatment with albumin-bound paclitaxel, oxaliplatin, tegafur,gimeracil and oteracil porassium capsules and sintilimab.

INTERVENTIONS:
Drug: Perioperative treatment with albumin-bound paclitaxel, oxaliplatin, tegafur,gimeracil and oteracil porassium capsules and sintilimab. — 1. Neoadjuvant therapy for 4 cycles: albumin-bound paclitaxel 150mg/m2, intravenously, d1, a course of treatment every 21 days; sintilimab 200mg, intravenously, d1, every 21 days; tegafur,gimeracil and oteracil porassium (by body surface area: BSA<1.25m2, 40mg; BSA≥1.25m2, <1.5m2, 50mg; BSA≥1.5m2,60mg), orally, twice a day, d1-14, every 21 days; oxaliplatin 85mg/m2, intravenously, d1, every 21 days.
  2. Radical surgical treatment should be performed within 4-6 weeks after the end of neoadjuvant therapy.
  3. Adjuvant therapy for 4 cycles: albumin-bound paclitaxel 125mg/m2, intravenously, d1, a course of treatment every 21 days; sintilimab 200mg, intravenously, d1, every 21 days; tegafur,gimeracil and oteracil porassium (by body surface area: BSA<1.25m2, 40mg; BSA≥1.25m2, <1.5m2, 50mg; BSA≥1.5m2,60mg), orally, twice a day, d1-14, every 21 days.

SUMMARY:
The goal of this clinical trial is to learn if treatment modality including albumin-bound paclitaxel, oxaliplatin, tegafur,gimeracil and oteracil porassium capsules (SOX) and sintilimab works to treat locally advanced HER2-negative hepatoid adenocarcinoma of stomach. It will also learn about the safety of this modality. The main aim it aims to achieve are:

* To evaluate the perioperative efficacy of albumin-bound paclitaxel combined with sintilimab and SOX in the treatment of locally advanced HER2-negative hepatoid adenocarcinoma of stomach
* To evaluate the safety and long-term benefits of albumin-bound paclitaxel combined with sintilimab and SOX regimens in perioperative treatment of locally advanced HER2-negative hepatoid adenocarcinoma of stomach

Participants will:

* Preoperative treatment with abumin-bound paclitaxel, SOX and sintilimab for 4 cycles
* Radical surgery after 4-6 weeks of the preoperative treatment
* Adjuvant treatment with albumin-bound paclitaxel, tegafur,gimeracil and oteracil porassium capsules and sintilimab for 4 cycles

ELIGIBILITY:
Inclusion Criteria:

* The histological type of gastric hepatoid adenocarcinoma was confirmed by pathological biopsy；
* HER2 negative (Immunohistochemistry: 0);
* Patients with clinical stage II-III;
* Those who are expected to complete R0 excision;
* ECOG score 0~1;
* Generally in good condition, perioperative treatment and surgical resection can be tolerated;
* Patients were enrolled voluntarily.

Exclusion Criteria:

* Combined with other malignant tumors (excluding thyroid papillary carcinoma, facial basal cell carcinoma and other low-grade malignant tumors); -Patients with obstruction, bleeding, etc. who need surgical intervention after evaluation by clinicians;
* dMMR/MSIH status；
* Received other anti-tumor therapy before enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-18 (Actual); Primary Completion 2027-09-20 (Estimated); Study Completion 2028-09-20 (Estimated)

PRIMARY OUTCOMES:
pathological complete response rate | within 10 days after surgery
  The proportion of subjects with node-negative lymph nodes and without residual viable tumor cells in the total number of subjects

SECONDARY OUTCOMES:
major pathological response rate | Within 10 days after surgery
  The proportion of subjects with surviving tumor cells ≤10% in total subjects; Time Frame: within 10 days after surgery
Objective response rate | From enrollment to surgery, assessed up to 3 months
  Proportion of patients who achieved pre-defined tumor volume reduction , including patients with complete response (CR) and partial response (PR).
Event-free survival | From date of enrollment until the date of first documented progression, recurrence or date of death from any cause, whichever came first, assessed up to 3 years
  From the start of treatment to the first occurrence of any of the following events: disease progression without surgical treatment, local or distant recurrence, death from any cause
Disease free survival | From date of surgery until the date of first documented recurrence or date of death from any cause, whichever came first, assessed up to 3 years
  It usually starts from the time when the patient receives treatment (such as surgery), and ends at the time when the disease recurs (such as tumor recurrence, metastasis) or when the patient dies for any reason
overall survival | From date of diagnosis until the date of death from any cause, assessed up to 3 years
  It refers to the period from when the patient is diagnosed until death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Jiafu Ji, MD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Peking University Cancer Hospital & Institute, Beijing, China